CLINICAL TRIAL: NCT00005395
Title: Honolulu Heart Program-Study of Stroke and Dementia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4303; R01HL054280 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-02

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Cerebrovascular Disorders; Dementia
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Cerebrovascular Disorders; Dementia

SUMMARY:
To clarify the relationship of the arterial lesions to aging, define the influence of the arterial changes on the development of stroke, brain infarction, and dementia, and provide a better understanding of vascular dementia.

DETAILED DESCRIPTION:
BACKGROUND:

Morphologic delineation of the arterial lesions will assist the use of experimental models to study molecular mechanisms underlying the lesions and the development of pharmacologic methods for controlling these mechanisms. Further examination of risk factors for the arterial lesions will indicate opportunities for prevention or modifying their evolution.

DESIGN NARRATIVE:

The study was based on data including risk factors and autopsy brain sections from deceased men from the Honolulu Heart Program. In this cohort, medial and intimal lesions of brain parenchymal arteries were significantly associated with brain infarction and three times more common in men dying of stroke than of non-cardiovascular causes. The specific aims of the study were 1) delineation of the morphologic characteristics of the brain parenchymal artery lesions, their regional anatomic distribution, and their relationship to changes in adjacent brain parenchyma and the degree of atherosclerosis in the major intracranial arteries; 2) characterization of the relationship in men between the arterial lesions and advancing age; 3) characterization in men over 60-65 years of age of the relationship of the arterial lesions to stroke, brain infarction or hemorrhage, and dementia; 4) identification of additional risk factors associated with the arterial lesions. The arterial lesions and adjacent brain parenchyma were examined with conventional histologic stains and immunohistochemical markers for specific cellular and extracellular components of the arterial wall. The prevalence and extent of each type of arterial lesion were determined at three anatomic sites. Baseline risk factors thought to be related to stroke and brain infarction were examined for association with the arterial lesions. Statistical tests of association were based on univariate and multivariate linear and logistic regression models controlled, when necessary, for age.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Nelson — Louisiana State University Medical Center

REFERENCES:
- [Background] Nelson JS. Alzheimer pathology in elderly patients with glioblastoma multiforme. Arch Pathol Lab Med. 2002 Dec;126(12):1515-7. doi: 10.5858/2002-126-1515-APIEPW. PMID 12456214
- [Background] Kehl F, Pagel PS, Krolikowski JG, Gu W, Toller W, Warltier DC, Kersten JR. Isoflurane does not produce a second window of preconditioning against myocardial infarction in vivo. Anesth Analg. 2002 Nov;95(5):1162-8, table of contents. doi: 10.1097/00000539-200211000-00006. PMID 12401584
- [Background] Abbott RD, White LR, Ross GW, Masaki KH, Curb JD, Petrovitch H. Walking and dementia in physically capable elderly men. JAMA. 2004 Sep 22;292(12):1447-53. doi: 10.1001/jama.292.12.1447. PMID 15383515